CLINICAL TRIAL: NCT04895397
Title: Modified Pectoral Nerve Block Versus Serratus Plane Block for Analgesia After Breast Cancer Surgeries
Brief Title: Modified Pectoral Nerve Block Versus Serratus Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Hussin Mohamed, principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: soh-Med-21-02-05
Record Dates: First submitted 2021-04-24; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A: (30 patients) modified pectoral nerve block will be done.
  Group B: (30 patients) serratus plane block will be done.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (30 patients) (Active Comparator): modified pectoral nerve block will be done.
  Interventions: Device: ultrasound guided Nerve Block procedure
- Group B: (30 patients) (Active Comparator): serratus plane block will be done.
  Interventions: Device: ultrasound guided Nerve Block procedure

INTERVENTIONS:
Device: ultrasound guided Nerve Block procedure — In group A patients, an ultrasound guided modified pectoral nerve block will be performed Under sterile conditions, US-guided PECSII block will be on the same side of surgery . The 6-13 MHz linear probe will be put transversely in the ipsilateral clavipectoral triangle - between the clavicle medially and above and the shoulder joint laterally.
  the needle will be advanced in an in-plane technique targeting the space in which the artery is located. Afterward, 10 mL of bupivacaine, 0.25%, will be injected.
  the needle will be advanced in-plane targeting the plane between the pectoralis minor muscle and serratus. Two mL of saline 0.9% will be injected; then, 10 mL of bupivacaine 0.25% will be injected.
  Group B: In SAPB Group, a US-guided serratus block will be done The ribs will be then counted, and when the 4th rib will be identified, the high-frequency probe will be put over it, in the mid-axillary line in a sagittal plane.

SUMMARY:
In PECSII or modified PECSI block, local anesthetic (LA) is injected between pectoralis major muscle (PMm) and pectoralis minor muscle (Pmm) to block lateral and medial pectoral nerves and between pectoralis minor muscle (Pmm) and serratus anterior muscle in the anterior axillary line to block the intercostal nerves II-VI (Blanco et al., 2012).

In Serratus anterior plane block (SAPB) local anesthetic (LA) is injected above the serratus muscle (between latissmus dorsi muscle and serratus muscle) or below the serratus muscle (between serratus muscle and 4th rib) in the mid-axillary line to block the intercostal nerves II-VI and spares the pectoral nerves (Blanco et al., 2013).

DETAILED DESCRIPTION:
One hour before induction of anesthesia 4ml blood sample will be taken from all patient to measure serum cortisol and serum endorphin level 2ml for each.

General anesthesia will be induced for all patients in both groups using the same protocol.

Anesthesia will be induced with propfol (2-3 mg/kg), IV rocuroniom (.5 - .8 mg/kg) to facilitate endotracheal intubation. Anesthesia will be maintained with isoflurane (1-2 mac) in 100% oxygen.

All patients will be intubated and mechanically ventilated using volume controlled positive pressure ventilation with a tidal volume of 6-8 ml/kg and an inspiratory to expiratory ratio of 1:2 targeting end tidal carbon dioxide tension around 35mmhg.

Basic monitoring for all patients include under pulse oximetry, non-invasive blood pressure, 5 lead electrocardiogram and end tidal carbon dioxide monitoring.

In group A patients, an ultrasound guided modified pectoral nerve block will be performed after induction of general anesthesia. Under sterile conditions, US-guided PECSII block will be on the same side of surgery with the patient lying in the supine position with the ipsilateral arm abducted and externally rotated, and the elbow flexed 90°. The 6-13 MHz linear probe will be put transversely in the ipsilateral clavipectoral triangle - between the clavicle medially and above and the shoulder joint laterally.

After identification of the Pectoralis major muscle, Pectoralis minor muscle and the plane in between, the probe will be tilted caudally to identify the pulsating pectoral branch of the thoracoacromial artery, if not identified, the probe will be moved 1-2 cm caudally and medially. In a caudal tilt, the artery will be easily identified in a biconvex space.

The skin at the point of entry was infiltrated using lidocaine 1%; then, the needle (disposable spinal needle, K-3 point type LUER-Lock HUB 22G) will be advanced in an in-plane technique targeting the space in which the artery is located. Two mL of saline 0.9% will be injected to confirm the location, produce hydro-dissection, and improve needle visualization. Afterward, 10 mL of bupivacaine, 0.25%, will be injected.

Then, the probe will be moved laterally and caudally towards the anterior axillary fold, parallel to the deltopectoral groove, until the serratus muscle appears underneath the Pectoralis minor muscle attached to the underlying ribs.

The 3rd, fourth ribs and the pleura will be then identified. After infiltration of the skin with lidocaine 1%, the needle will be advanced in-plane targeting the plane between the pectoralis minor muscle and serratus. Two mL of saline 0.9% will be injected; then, 10 mL of bupivacaine 0.25% will be injected.

Group B: In SAPB Group, a US-guided serratus block will be done with the patient in the lateral position, with the side of the surgical side up and the upper limb hanging over the patient's head. The ribs will be then counted, and when the 4th rib will be identified, the high-frequency probe will be put over it, in the mid-axillary line in a sagittal plane.

The ribs, pleura, and overlying serratus muscle will be identified, and the needle will be advanced cephalad in-plane until the tip touched the 4th rib. Afterward, 2 mL saline 0.9% will be injected; then, 20 mL of bupivacaine 0.25% will be injected in the plane between the serratus and the 4th rib.

At the end of the surgery, the muscle relaxant will be reversed using neostigmine (0.04 mg/kg) and atropine (0.01 mg/kg). After fully awake extubation, all patients will be transferred to the post-anesthesia care unit (PACU).

Two hour post-operative 4ml blood sample will be taken from all patients to measure serum cortisol and serum endorphin level 2ml for each.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer surgery.
* Age 20 to 60 years.
* Female patients.
* At least 24 hours post-operative hospital admission.
* ASA (American society of anesthesiologist) physical status classification system І to Ш.

Exclusion Criteria:

* • Morbid obesity (body mass index > 40).

  * Impossibility of anatomical structures identification by ultrasound in a satisfactory way (there can be no distinction in the interfacial plan between serratus and pectoral muscle).
  * Opioids treatment before surgery or substance abuse.
  * Sepsis and/or infection at the puncture site.
  * Hemostasis disorders.
  * Allergy to any of the drugs used in the study.
  * Less than 24 hours postoperative hospital admission.
  * Inability to communicate with the patient.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
assess analgesic effect of nerve block | 24hour post-operative
  We assess the analgesic effect by VAS ( visual analogue scale )

CONTACTS AND LOCATIONS:
Overall Officials: mohammed hussein, lecturer, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No